CLINICAL TRIAL: NCT03399825
Title: Investigation of Vascular Pathology in Eye Diseases Using Optical Coherence Tomography Angiography (OCT-A) in Children (≥ 6 <14 Years of Age)
Brief Title: Optical Coherence Tomography Angiography (OCT-A) in Children (≥ 6 <14 Years of Age)
Acronym: OCTAC
Status: Withdrawn | Type: Observational
Why Stopped: administrative hurdles
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: OCTA children
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Retinopathy of Prematurity; Diabetic Retinopathy
MeSH Terms: conditions — Retinopathy of Prematurity; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: Children without eye disease
  Interventions: Device: OCT-A
- Retinopathy of prematurity (ROP): Previously preterm children with a history of ROP
  Interventions: Device: OCT-A
- Diabetic retinopathy: Children with diabetes
  Interventions: Device: OCT-A

INTERVENTIONS:
Device: OCT-A — optical coherence tomography angiography
  Imaging with optical coherence tomography angiography

SUMMARY:
Comparison of OCTA to conventional imaging modalities for the diagnosis of eye diseases in children

DETAILED DESCRIPTION:
Optical coherence tomography angiography (OCTA) is a new non-invasive imaging technique that employs motion contrast imaging to high-resolution volumetric blood flow information. OCTA compares the decorrelation signal between sequential OCT b-scans taken at precisely the same cross-section in order to construct a map of blood flow. At present, level 1 evidence of the technology's clinical applications doesn't exist. The investigators plan to compare OCTA as an imaging modality to conventional imaging modalities used in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Patients (children ≥ 6 <14 years of age) from the Childrens Hospital, University Hospital Bern requiring routine internal medical check-up for the diagnosis of diabetes or children attending routine eye exams at the department of ophthalmology, who are willing to participate in the study, and whos parents are willing to sign informed consent on behalf of their child.
* Patients need to be at least 6 years of age (but younger than 14 years) 6 years of age or younger

Exclusion Criteria:

* Patients (children) who are not willing or able to participate, or potential participant's parents who are not willing to sign informed consent on behalf of their child.
* Patients younger than 6 years of age or 14 years or older.
* Patients (children) with epilepsy

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants with a history of clinically diagnosed retinal diseases and healthy individuals undergoing ophthalmic Imaging in Routine clinical practice will be included
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the sensitivity and specificity of OCTA | 2 years
  The primary objective of this observational study is to evaluate the sensitivity and specificity to diagnose vascular abnormalities with OCTA compared to conventional imaging methods. The main parameter that will be assessed is area of nonperfusion of the retina. The incidence (binary) of nonperfusion areas will be assessed in OCTA and compared to conventional imaging methods such as fluorescein angiography.